CLINICAL TRIAL: NCT03583463
Title: A Prospective Non-InterventionaL Study To EXplore the Real-Life MAnagement Of Postmenopausal womeN With Hormone Receptor- Positive, Human EpiDermal Growth Factor Receptor 2-Negative Locally Advanced/ MetastatIc BreAst Cancer In Egypt
Brief Title: ALEXANDRIA Study Egypt
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00138
Record Dates: First submitted 2018-06-27; First posted 2018-07-11 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Device: No

SUMMARY:
Breast Cancer (BC) is one of the most frequent cancers in women and is the most frequent cause of death in the female population. It represents 18% of all female cancers in the world.1 The incidence varies in different populations with almost half of the cases having their origin in North America and Western Europe. In Egypt, according to the National Population-Based Cancer Registry published in 2014, BC was the most frequent cancer among females representing 32% of all female cancers2 Metastatic disease occurs in approximately 20-50% of patients with early BC history and in 6-10% of newly diagnosed BC cases.3 Since patients with metastatic BC form a heterogeneous population, treatment recommendations ought to be made on an individual basis, considering hormone receptor (HR) and human epidermal growth factor receptor 2 (HER2) status, metastasis-free interval (MFI), response to and cumulative doses of previous therapy, location and extent of metastases and symptoms 4,5.

Two thirds of BC patients have HR-positive (HR+) tumors 6, for whom endocrine therapy (ET) is the preferred initial treatment for metastatic disease as recommended in the treatment guidelines, even in the presence of visceral metastases 4, 6, 7. The use of ET is supported by data showing a therapeutic benefit with less toxicity and better quality of life in comparison to chemotherapy (CT) 5,8,9. Nevertheless, it is generally thought that CT is associated with greater and earlier tumor response, especially in the case of high burden of disease. For patients with hormone receptor-positive and HER2+ disease CT plus HER2-targeted therapy was strongly recommended, except for highly selected cases for whom clinicians may offer ET 10. On the contrary, for women with hormone receptor-positive HER2-negative disease who are the scope of this study the question of whether to use CT or ET as first-line treatment for metastatic BC remains, to date, partially unresolved.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study specific procedures
2. Post-menopausal women (Defined as a woman who have experienced at least 12 consecutive months without menstruation, who had undergone bilateral ovariectomy or who has menopausal levels of serum Estradiol and FSH.)
3. Hormone receptor positive, HER2 negative locally advanced or metastatic breast cancer.
4. Patients with either de novo metastatic disease who had not received any prior treatment or those who progressed during or after previous adjuvant endocrine treatment for early breast cancer.
5. Hormone sensitive patients (per the ABC2 guidelines published in Annals of Oncology 00: 1-18, 2014, defined as relapse while on adjuvant ET but after the first 2 years, or a relapse after/within 12 months of completing adjuvant ET. Patients with ER+ de novo metastatic disease are also considered hormone sensitive patients)
6. Patients have already been prescribed treatment with ET either as monotherapy or in combination or physician's choice of a standard of care chemotherapy within the previous 90 days prior to their enrolment.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous inclusion in the present study
3. Current enrollment and/or participation in another clinical study during the last 90 days.
4. Presence of visceral crisis.
5. Failure to meet any of the inclusion criteria.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with ER positive, HER-2 negative locally advanced/ metastatic breast cancer, who either progressed during or after adjuvant endocrine therapy for early breast cancer or those presenting with de novo metastatic disease who had not received prior endocrine therapy. Patients should have already been prescribed first line treatment for their locally advanced/ metastatic breast cancer as per routine clinical practice prior to their enrolment in the study. Their participation in the study should in no way impact the treatment and care that they receive.
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with ER positive, HER2 negative locally advanced or metastatic breast cancer assigned to each treatment modality used as the first line of treatment. | 18 Months
  Proportion of patients with ER positive, HER2 negative locally advanced or metastatic breast cancer assigned to each treatment modality used as the first line of treatment.
Characteristics of patients in each treatment modality according to their histologic diagnosis, Hormone sensitivity, visceral vs non-visceral disease proportion, reason for selecting the treatment. | 18 Months
  Characteristics of patients in each treatment modality according to their histologic diagnosis, Hormone sensitivity, visceral vs non-visceral disease proportion, reason for selecting the treatment.

SECONDARY OUTCOMES:
Progression-free survival of patients receiving first line treatment for ER positive, HER2 negative locally advanced or metastatic breast cancer, for all patients. | 18 Months
  Progression-free survival of patients receiving first line treatment for ER positive, HER2 negative locally advanced or metastatic breast cancer, for all patients.
Response Rate (RR) of patients receiving first line treatment for ER positive, HER2 negative locally advanced or metastatic breast cancer. | 18 Months
  Response Rate (RR) of patients receiving first line treatment for ER positive, HER2 negative locally advanced or metastatic breast cancer.
Proportions of patients on each second line treatment modality in patients diagnosed with ER positive, HER2 negative locally advanced or metastatic breast cancer. | 18 Months
  Proportions of patients on each second line treatment modality (subsequent therapy following progression on first line treatment described in primary outcome variable) in patients diagnosed with ER positive, HER2 negative locally advanced or metastatic breast cancer.

CONTACTS AND LOCATIONS:
Locations (8):
- Egypt (8):
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, El Gharbia
  - Research Site, El Menofia
  - Research Site, Gharbia
  - Research Site, Giza
  - Research Site, Luxur
  - Research Site, Zagazig

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00138&attachmentIdentifier=871f3022-a600-4bd8-a27d-914b53f6db4a&fileName=CSR_Synopsis_ALEXANDRIA_(D133FR00138)_Redacted.pdf&versionIdentifier=